CLINICAL TRIAL: NCT05049850
Title: An Open Label, Phase II Study to Investigate DSA Rebound in Patients With a Positive Crossmatch, Made Transplantable With Imlifidase
Brief Title: A Study to Investigate DSA Rebound in Patients Treated With Imlifidase Prior to Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision, not due to any safety reason
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-HMedIdeS-16
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Kidney Transplantation in Highly Sensitized Patients
Keywords: Highly sensitized; Kidney transplantation; Renal transplantation
MeSH Terms: interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imlifidase (Experimental): Imlifidase is administered intravenously as one dose of 0.25 mg/kg over 15 minutes within the 24-hour period prior to transplantation. (A second dose may be given if the crossmatch test at 4 hours after the first dose remains positive.)
  Interventions: Drug: Imlifidase

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly specific for IgG.
  Other Names: IdeS, HMED-IdeS

SUMMARY:
The purpose of this study is to assess whether imlifidase in combination with bortezomib, belatacept, rituximab and IVIg can suppress donor specific antibodies (DSA) and the occurrence of antibody-mediated rejection (AMR) in highly sensitized patients with chronic kidney disease with a positive crossmatch towards their living donor during a period of 3 months from transplantation.

DETAILED DESCRIPTION:
Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly specific for IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG. Clinical studies with imlifidase have demonstrated that the treatment enables transplantation in patients otherwise highly unlikely to be transplanted, by converting a positive crossmatch to a negative.

However, as with other desensitization methods, DSA tend to reappear within weeks after treatment and transplantation, which may cause AMR and increased risk of graft loss. In this study, treatment with imlifidase in combination with approved drugs that prevent or suppress DSA rebound by targeting antibody-producing plasma-cells and their B-cell precursors is suggested. These drugs include (i) bortezomib, a proteasome inhibitor which has activity against mature plasma cells, the source of DSA, (ii) belatacept, a fusion protein which is crucial in blocking T-cell co-stimulation and which is effective in reducing de novo DSA generation in humans, (iii) rituximab, an anti-CD20 monoclonal antibody that targets B-cells and which is an immunomodulatory agent, and (iv) intravenous immunoglobulin (IVIg) which is commonly used in desensitization regimens and for the treatment of AMR.

After being informed about the study and potential risks, all patients giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry. Patients who meet the eligibility requirements will then start treatment with belatacept and bortezomib about 3 weeks prior to the imlifidase infusion and transplantation. Rituximab will be initiated 8 days after transplantation and IVIg 10 days after transplantation. Induction and maintenance immunosuppression will also be administered. The patients will be hospitalized for approximately 2 weeks following transplantation and after that 9 follow-up visits to the clinic will take place up to 6 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent obtained before any trial-related procedures
* Male or female age 18 to 70 years at the time of screening
* Highly sensitized patients registered on the UNOS waiting list for kidney transplantation, with either of the following:

  * cPRA ≥ 99.9%
  * cPRA ≥ 98% and have been in kidney paired donation or kidney paired exchange programs for at least 1 year
* A positive crossmatch towards a living donor
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Previous treatment with imlifidase
* Previous high dose IVIg treatment (2 g/kg) within 28 days prior to imlifidase treatment
* Breast-feeding or pregnancy
* Women of child-bearing potential not willing or able to practice FDA-approved forms of contraception. Two medically acceptable methods of highly effective contraception must be used for the duration of the study (e.g. oral, transdermal, intravaginal, injectable or implantable contraceptive; intrauterine device; intrauterine hormone-releasing system; vasectomized partner; bilateral tubal occlusion; or double-barrier method). For a woman to be considered postmenopausal this ascertainment must be made according to medical records and clinical history and may be aided by measurement of elevated postmenopausal serum gonadotropin levels (FSH).
* ABO blood group incompatible transplantations (A2 and A2B kidneys will not be accepted for B recipients)
* Positive serology for HIV
* Clinical signs of HBV, HCV, CMV, or EBV infection
* EBV seronegative or with unknown EBV serostatus
* Positive SARS-CoV-2 tests at any time point from screening to transplantation
* Active tuberculosis
* Ongoing serious infections as judged by the investigator
* Severe other conditions requiring treatment and close monitoring e.g. cardiac failure ≥ grade 4 (New York Heart Association), unstable coronary disease or oxygen dependent respiratory disease
* A history of a proven hypercoagulable condition
* Present, or history of, thrombotic thrombocytopenic purpura (TTP) or known familial history of TTP
* Intake of investigational drugs (other than imlifidase) within 5 half-lives
* Contemporaneous participation in a medical device study
* Known allergy/sensitivity (except local reactions) to imlifidase or to any drug (or the excipients) specified in the protocol
* Known mental incapacity or language barriers precluding adequate understanding of the Informed Consent information and the trial activities
* Inability by the judgement of the investigator to participate in the trial for any other reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (1):
- NYU Langone Health Transplant Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Sponsor decided to prematurely terminate the trial after 3 of the 12 patients had been treated and transplanted in the trial due to prioritization of internal resources. This decision was unrelated to either safety or efficacy, no safety issues were raised during the conduct of the trial.
Period: Overall Study
Arm/Group | Imlifidase
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With DSA Rebound
Description: The recurrence of DSA may cause AMR and increased risk of graft loss. Due to the early termination of the trial the primary endpoint was assessed as the incidence of DSA rebound of either immunodominant or total DSA to a mean fluorescence intensity (MFI) level that was ≥50% of the pre-imlifidase value up to 3 months after transplantation (trial day 91).
Time Frame: Up to 3 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Proportion of Patients With Kidney Biopsy Proven AMR
Description: The standardized international Banff classification 2019 for assessment of renal allograft biopsies will be used to assess AMRs reported from the study based on for cause and protocol biopsies.
Time Frame: Up to 6 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Proportion of Patient With DSA Rebound
Description: See description to primary outcome measure
Time Frame: Up to 6 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Proportion of Patients With Negative FCXM
Description: Imlifidase is highly efficacious in converting a positive crossmatch to a negative
Time Frame: Up to 24 hours after imlifidase treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Levels of DSA
Description: Analysis of DSAs before and after imlifidase will be done. The mean fluorescence intensity (MFI) will be presented for the individual patients' DSAs.
Time Frame: Within 4 hours before imlifidase until Day 181
Population: Only 2 of 3 patients had data for DSA collected at the Day 181 timepoint, for patient 2 data from an unscheduled visit at day 139 is presented.
Measure: Number; unit: MFI
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
MFI
  Patient 1, pre-dose: number analyzed (Participants) | 1
  Patient 1, pre-dose | 22311
  Patient 1, Day 181: number analyzed (Participants) | 1
  Patient 1, Day 181 | 8619
  Patient 2, pre-dose: number analyzed (Participants) | 1
  Patient 2, pre-dose | 8526
  Patient 2, Day 139: number analyzed (Participants) | 1
  Patient 2, Day 139 | 2172
  Patient 3, pre-dose: number analyzed (Participants) | 1
  Patient 3, pre-dose | 9994
  Patient 3, Day 181: number analyzed (Participants) | 1
  Patient 3, Day 181 | 149

6. Secondary Outcome: Levels of Complement Binding (C1q) DSA
Description: Analysis of C1q DSAs before and after imlifidase will be done. The mean fluorescence intensity (MFI) will be presented for the individual patients' C1q DSAs.
Time Frame: Within 4 hours before imlifidase until Day 181
Population: Samples for assessment of DSA, including Cq1 DSA, were collected. However, the central laboratory assigned to Cq1 DSA analyzes was never activated due to the premature trial termination, hence analysis of Cq1 DSA was not performed.
Arm/Group | Imlifidase
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Graft Survival
Description: Graft survival will be summarized by end of trial.
Time Frame: 6 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 3

8. Secondary Outcome: Patients Survival
Description: Patient survival will be summarized by end of trial.
Time Frame: 6 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 3

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety is assessed as type, frequency and intensity of adverse events (AEs)/serious adverse events (SAEs) including clinically relevant changes in clinical laboratory tests, vital signs and ECG)
Time Frame: Up to 6 months after transplantation
Population: Results for adverse events is presented in the section Reported Adverse Events.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
Participants | 3

10. Secondary Outcome: Kidney Function Assessed by Creatinine
Description: P-creatinine is a measure of kidney function.
Time Frame: Up to 6 months after transplantation
Measure: Median (Full Range); unit: μmol/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
μmol/L
  Pre-dose | 506 [305 to 682]
  Day 181 | 180 [91 to 184]

11. Secondary Outcome: Kidney Function Assessed by Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated glomerular filtration rate (eGFR) is a measure of kidney function. eGFR will be calculated as described by the modification of diet in renal disease (MDRD) equation.
  eGFR for a kidney with normal function is 90 mL/min/1.73m2. Kidney disease is characterized by a decreased eGFR value.
Time Frame: Up to 6 months after transplantation
Measure: Median (Full Range); unit: mL/min/1.73m2
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
mL/min/1.73m2
  Pre-dose | 11 [6 to 14]
  Day 181 | 35 [26 to 60]

12. Secondary Outcome: Kidney Function Assessed by Protein/Creatinine Ratio in Urine
Description: The protein/creatinine ratio in urine is a measure of kidney function. Will be measured unless patients are anuric.
Time Frame: Up to 6 months after transplantation
Population: Only 2 of the 3 patients had data collected at the Day 181 timepoint.
Measure: Median (Full Range); unit: mg/g
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
mg/g
  24h post-dose | 2158 [1900 to 120025]
  Day 181: number analyzed (Participants) | 2
  Day 181 | 1233 [470 to 1996]

13. Secondary Outcome: Imlifidase Pharmacokinetics (AUC)
Description: AUC = Area under the imlifidase plasma concentration versus time curve
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: h×μg/mL
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
h×μg/mL | 71.9 [65.6 to 119]

14. Secondary Outcome: Imlifidase Pharmacokinetics (Cmax)
Description: Cmax = Maximum observed plasma concentration of imlifidase following dosing
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
μg/mL | 3.70 [3.20 to 4.10]

15. Secondary Outcome: Imlifidase Pharmacokinetics (Tmax)
Description: tmax = Time point for maximum observed plasma concentration of imlifidase following dosing
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: h
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
h | 1.13 [1.00 to 1.25]

16. Secondary Outcome: Imlifidase Pharmacokinetics (t1/2)
Description: t1/2 = Terminal half-life of imlifidase, the time taken for concentration of imlifidase to decrease from its maximum concentration (Cmax) to half of Cmax in the blood plasma.
  t1/2 alpha = alpha phase (distribution/elimination) half-life, an initial phase of rapid decrease in plasma concentration.
  t1/2 beta = beta phase (elimination) half-life, a phase of gradual decrease in plasma concentration after the alpha phase.
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: h
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
h
  t1/2 alpha | 6.40 [1.05 to 9.29]
  t1/2 beta | 28.3 [26.7 to 37.2]

17. Secondary Outcome: Imlifidase Pharmacokinetics (CL)
Description: CL = Clearance of imlifidase
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: mL/h/kg
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
mL/h/kg | 3.48 [2.11 to 3.81]

18. Secondary Outcome: Imlifidase Pharmacokinetics (Vz)
Description: Vz = Apparent volume of distribution during terminal phase
Time Frame: Within 4 hours before imlifidase dose until Day 15
Measure: Median (Full Range); unit: L/kg
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
L/kg | 0.142 [0.081 to 0.205]

19. Secondary Outcome: Pharmacodynamics
Description: Concentration of IgG in patient serum will be measured. Scoring of IgG fragments will be done.
Time Frame: Within 4 hours before imlifidase dose until Day 10
Measure: Median (Full Range); unit: g/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
g/L
  Pre-dose | 11.6 [5.2 to 15.7]
  Day 10 | 1.0 [0.6 to 3.4]

20. Secondary Outcome: Anti-drug Antibodies (ADA) Levels
Description: Immunogenicity towards imlifidase will be assessed by the measurement of ADA levels in patient serum using a customized ImmunoCAP analysis.
Time Frame: Up to 6 months after imlifidase
Measure: Median (Full Range); unit: mg/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
mg/L
  Pre-dose | 4.1 [2.4 to 82.9]
  Day 181 | 20.5 [13.7 to 30.2]

21. Secondary Outcome: Change in Patient-reported Life Participation, as Measured PROMIS-SF-8a
Description: The PROMIS Social Health domain "Ability to participate in social roles & activities PROMIS-SF-8" will be used as a measure of the patients' health related quality of life.
Time Frame: At screening and Day 181
Population: PROMIS-SF-8 sores are calculate using the PROMIS® Short Form v2.0-Ability to Participate in Social Roles and Activities 8a scoring manual. The total scale raw score was translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10, i.e. a T-score of 40 is one SD below the mean. The lowest possible T-score is 25.9 and the highest possible score is 65.4, a higher score means a better outcome.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 3
score on a scale
  Screening | 53.6 [44 to 54.6]
  Day 181 | 65.4 [60.2 to 65.4]

ADVERSE EVENTS:
Time Frame: AEs were collected on the AE CRF for each patient, from the time of signing of the informed consent and throughout the trial including the follow-up period. 35 Days in screening phase plus 181 Days in trial, a total of 216 Days.
Arm/Group | Imlifidase
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Wound evisceration (Infections and infestations) | 1 (1)
Donor specific antibody present (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Delayed graft function (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT05049850/Prot_SAP_001.pdf